CLINICAL TRIAL: NCT00661843
Title: A Mixed Design, With Wait List Control Crossover to Intervention, Clinical Trial of Integrated Yoga Style Practice Intervention for Improving Sleep and Quality of Life in the Elderly Population
Brief Title: A Study of Yoga for Treating Geriatric Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Collaborators: KTH Royal Institute of Technology (Other); The Australia-Israel Scientific Exchange Foundation (AISEF) (Other); Israel Yoga Teachers Association (Unknown)
Responsible Party: Dr. Clement Cahan, head of the Sleep Lab, Shaare Zedek Medical Center, Shaare Zedek Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SZMCSL0001
Record Dates: First submitted 2008-04-16; First posted 2008-04-18 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2010-08

CONDITIONS: Primary Geriatric Insomnia; Sleep Initiation and Maintenance Disorders
Keywords: insomnia; geriatric; yoga; sleep; electrocardiogram
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Intervention group: Intervention constitutes of 2 supervised yoga classes per week incorporating gentle Yoga postures, relaxation and meditation sequences In addition: daily home based sessions of yogic relaxation and meditation using a pre-recorded audio CD
  Interventions: Other: Integrated Yoga style practice
- 2 (No Intervention): Control in waiting to be crossed over after control phase completed. Participants of this group studied using same objective and subjective outcome measures.

INTERVENTIONS:
Other: Integrated Yoga style practice — Intervention constitutes of 2 supervised yoga style classes per week incorporating gentle postures,relaxation and meditation sequences. In addition daily home based sessions of yogic relaxation, and meditation a an audio CD
  Arms: 1

SUMMARY:
Insomnia is common in the elderly population and is associated with increased health problems, reduced quality of life and greater use of sleep inducing drugs. This research aims to examine the effectiveness of Yoga practice to treat insomnia in elderly people, determine the ability to enhance their quality of life and determine if it is suitable to western culture and conditions.

DETAILED DESCRIPTION:
Introduction: Geriatric insomnia is prevalent, reducing life quality, diminishing cognition and increasing risk of accidents and mortality. Treatment with sedative-hypnotic drugs has limited effectiveness and further increases the risk of accidents and falls. Yoga has been shown to increase well-being in the elderly.

Hypotheses

1. Integrated yoga style practice can improve sleep quality/quantity
2. Integrated yoga style practice can improve quality of life.

Objectives:

1. Examine effectiveness of yoga for insomnia and reduction in use of hypnotics/relaxants in the elderly;
2. Determine whether yoga enhances quality of life in the elderly; and 3. Determine whether yoga is suitable for elderly in western culture(s).

Methods:

A mixed design crossover controlled trial (n =74, age range 60-87, M = 74.4, SD = 7.1) with 2 weekly classes incorporating physical and meditative yoga, and daily home practice of meditative yoga for 12 weeks. Measures included self-reported assessment of sleep quality (Sleep Logs, KSS, ESS, PSQI, MAPS), mood states (DASS, POMS), general health (SF-36) and mobile objective home sleep studies.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older
* Independent, self mobile
* Suffering from light to severe primary insomnia

Exclusion Criteria:

* Age less than 60 years
* Currently or in the past engaged in regular yoga practice
* Suffering from any physical or mental health condition or disability which may affect sleep, or for which Yoga practice is counter indicated or may lead to health risks or complications.
* Suffering from co-morbid insomnia in conjunction with another condition clearly salient to sleep disturbance.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2008-05; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Subjective sleep and life quality assessment using standard questionnaires and sleep logs | 24 weeks
  all measures taken at baseline and post intervention for all participants participant who crossed over measured pre and post control phase and post intervention phase
Objective home based sleep studies using | 24 weeks
  objective sleep studies using embletta mobile sleep recording system in conjunction with the HPC1000 sleep analysis system.
  all measures taken pre and post intervention. Participants who crossed over measured pre control, post control and post intervention phases

CONTACTS AND LOCATIONS:
Overall Officials: Anda Baharav, MD, Study Chair — Shaare Zedek Medical Center; Jonathan Halpern, M.Sc., Study Chair — Royal Melbourne Institue of Technology University; Clement Cahan, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Sleep Lab, Jerusalem, Israel, Israel